CLINICAL TRIAL: NCT04215952
Title: Optimizing and Understanding Semantic Feature Analysis Treatment for Aphasia: A Randomized Controlled Comparative Effectiveness Trial
Brief Title: Semantic Feature Analysis Treatment for Aphasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00003086
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Aphasia
Keywords: Anomia; Semantic Feature Analysis
MeSH Terms: conditions — Aphasia; Anomia

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of two treatment conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Administration and scoring of all primary and secondary outcome measures will be carried out by a speech pathologist on study staff who (1) is not the treating clinician for the participant being assessed, and (2) is blind to the group assignment of the participant being assessed. Because SFA is a behavioral intervention, it will not be possible to blind the treating clinician to group assignment. It will also be impossible to definitively blind participants to their group assignment. However, we will not formally disclose to participants the group to which they have been assigned, and in the informed consent process, we will describe the conditions only in relative terms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SFA Experimental Intervention (Experimental): A modified version of Semantic Feature Analysis will be administered.
  Interventions: Behavioral: Semantic Feature Analysis Treatment
- SFA Active Comparator Intervention (Active Comparator): A standard version of Semantic Feature Analysis will be administered.
  Interventions: Behavioral: Semantic Feature Analysis Treatment

INTERVENTIONS:
Behavioral: Semantic Feature Analysis Treatment — On each treatment trial, the clinician will show the participant with aphasia a pictured object and ask them to name it. The clinician will then guide the participant in verbally generating semantic features for the target, using a chart that specifies five kinds of features: group, use/action, properties, location, and personal associations. When the participant cannot generate a given feature, cueing or other assistance will be provided. After feature generation, the clinician will ask the participant to name the picture again and provide cueing if needed. The clinician will then review the generated features and ask the participant to name the item once more, with cueing if needed. Finally, the clinician will ask the participant to say a sentence containing the target word and provide cueing if needed. Treatment will then proceed to the next item. Participants will receive approximately 20 hours of treatment on each of three 10-item lists, for a total of 60 hours of treatment.
  Other Names: Semantically Oriented Naming Treatment

SUMMARY:
This randomized controlled comparative effectiveness study examines manipulation of a key component of an established and efficacious treatment for naming impairments in aphasia, along with cognitive and brain correlates of treatment success. Study participants will be randomly assigned to one of two treatment conditions comparing two different versions of Semantic Feature Analysis treatment. Their performance on standardized and study-specific measures will be used to determine which version of the treatment provides superior outcomes, and measures of automatic language processing and functional brain imaging will also be used to identify the underlying neurocognitive mechanisms associated with positive treatment response.

DETAILED DESCRIPTION:
This randomized comparative effectiveness trial examines whether active manipulation of a key component of semantic feature analysis (SFA) treatment for word-finding difficulty in aphasia improves outcomes. 40 study participants will be recruited and randomized to receive one of the two versions of the treatment. The total treatment time will be equated in the two conditions.

Study participants will be housed locally at the Pittsburgh site at no cost and will be eligible to receive reimbursement for travel expenses. During the five-week treatment phase of the study, participants will receive 60 hours of SFA treatment with pre- and post-treatment assessment of their ability to name pictures of treated and untreated, semantically related nouns. Other secondary outcomes, including measures of connected speech and patient-reported communication ability will also be collected. In order to address unresolved questions about the underlying cognitive and neural mechanisms of SFA, participants will also receive concurrent pre- and post-treatment assessment of automatic word processing ability using eye-tracking methods and functional magnetic resonance imaging (fMRI). Participants will also be asked to return to Pittsburgh for two days approximately 2-3 months later for follow-up language, eye-tracking, and fMRI testing.

The language testing results will be used to determine which version of SFA treatment optimizes outcomes. The eye-tracking results will be used to infer whether SFA's positive effects can be attributed to improved activation of lexical-semantic representations, improved ability to inhibit competing representations, or both. The fMRI results will be used to identify the brain networks and activation changes associated with changes in naming ability resulting from SFA. This study will provide theoretically and clinically relevant information about how aphasia treatment should be delivered and the neurocognitive mechanisms underlying its effects.

ELIGIBILITY:
Inclusion Criteria:

* 6 months post-onset of aphasia due to unilateral left-hemisphere (LH) stroke
* Independent in activities of daily living (ADLs) necessary to live in community-based housing or available caregiver to assist with ADLs
* Medically stable and able to tolerate intensive treatment schedule (e.g. no uncontrolled seizures, difficulty breathing, frequent migraines)
* English as a first language
* No participation in any other speech-language treatment during this study, including follow-up period
* Sufficient auditory comprehension abilities demonstrated during screening
* Sufficient naming impairment exhibited during screening

Exclusion Criteria:

* Right Hemisphere stroke
* Neurological disease other than stroke
* Significant psychiatric disorder
* Severe motor speech disorder
* Active substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Confrontation Naming | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in naming accuracy on 30 treated pictured object nouns and 30 untreated pictured object nouns semantically related to the treated items.

SECONDARY OUTCOMES:
Nicholas and Brookshire Picture Descriptions | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in the number of correct information units produced during connected speech in response to the stimuli and procedures described by Nicholas and Brookshire (1993) and Brookshire & Nicholas (1994).
Aphasia Communication Outcome Measure (ACOM) | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in ACOM T-scores derived from the scoring model described by Hula and colleagues (2015). Higher scores on this scale indicate better self-reported communicative functioning. The scale was constructed such that the average score is 50 and the standard deviation is 10 points. The minimum possible score is 15 and the maximum possible score is 85.
Visual World Paradigm | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in the mean proportions of fixations to the target and to the related competitor (compared to unrelated distractor images), averaged across trials.
Functional MRI | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Changes in task-related blood oxygen level dependent (BOLD) activation, and task-related and resting state functional connectivity
Comprehensive Aphasia Test | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in the Modality Mean T-Score computed from the following six modality subtests: Spoken Language Comprehension, Written Language Comprehension, Repetition, Naming, Reading, and Writing.
Philadelphia Naming Test (PNT) | (1) 1 week prior to intervention; (2) immediately prior to intervention; (3) 1-2 days post intervention (4) 8 to 12 weeks post intervention
  Change in PNT score estimates derived from the item response theory model described by Fergadiotis, Kellough, & Hula (2015). Scores will be scaled such that the expected average score among persons with aphasia is 50 and the standard deviation is 10, with minimum and maximum possible scores of approximately 20 and 80, respectively. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: William D Hula, Ph.D., Principal Investigator — VA Pittsburgh Healthcare System; Patrick J Doyle, Ph.D., Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Brookshire RH, Nicholas LE. Speech sample size and test-retest stability of connected speech measures for adults with aphasia. J Speech Hear Res. 1994 Apr;37(2):399-407. doi: 10.1044/jshr.3702.399. PMID 8028321
- [Background] Fergadiotis G, Kellough S, Hula WD. Item Response Theory Modeling of the Philadelphia Naming Test. J Speech Lang Hear Res. 2015 Jun 1;58(3):865-877. doi: 10.1044/2015_JSLHR-L-14-0249. PMID 25813461
- [Background] Hula WD, Doyle PJ, Stone CA, Austermann Hula SN, Kellough S, Wambaugh JL, Ross KB, Schumacher JG, St Jacque A. The Aphasia Communication Outcome Measure (ACOM): Dimensionality, Item Bank Calibration, and Initial Validation. J Speech Lang Hear Res. 2015 Jun;58(3):906-19. doi: 10.1044/2015_JSLHR-L-14-0235. PMID 25812178